CLINICAL TRIAL: NCT04119466
Title: Stabilizing Training Effects in Relation With Progression Level in Young Degenerative Disc Disease Individuals
Brief Title: Stabilizing Training in Degenerative Disc Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Błażej Cieślik, Research Assistant, Wroclaw University of Health and Sport Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MED23/2019
Record Dates: First submitted 2019-10-06; First posted 2019-10-08 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Degenerative Disc Disease; Protrusion; Extrusion of Migrated Disc; Hernia
Keywords: degenerative disc disease; stabilizing training; protrusion; extrusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Hernia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protrusion Group (Experimental): 20 session of stabilizing training based on the principles developed by Richardson over four weeks.
  Interventions: Behavioral: Stabilizing training
- Extrusion Group (Experimental): 20 session of stabilizing training based on the principles developed by Richardson over four weeks.
  Interventions: Behavioral: Stabilizing training

INTERVENTIONS:
Behavioral: Stabilizing training — The training will include the activation of the lumbar multifidus muscle (m. multifudus) and the transverse abdominal muscle (m. transversus abdominis). The performance of the individual stages of the training will be based on Richardson's methodology. One session will comprise 4 sets in which the patient will be asked to do pelvic tilts (draw-in) with simultaneous full exhalation, thus activating the aforementioned muscle groups in different positions: a) prone b) supine with lower extremities flexed c) quadruped d) standing back to the wall. The subjects will perform 3 series consisting of 10 repeats, each of which will last ca. 10 seconds.

SUMMARY:
This study evaluates efficacy of stabilizing training of deep core muscles in the lumbar spine in degenerative disc disease subjects, considering the progression level of degenerative disc disease: protrusion or extrusion.

DETAILED DESCRIPTION:
Degenerative disc disease (DDD) is one of the causes of low back pain, and contributes to increasing the socio-economic problem. Depending on the reason for the dysfunction, various classifications describing the level of advancement are used. Literature on the subject commonly uses the division into protrusion and extrusion of the intervertebral disc, as approved by the American Society of Neuroradiology.

Stabilizing training is one of the forms of conservative treatment of lumbar pain, alongside manual treatment or techniques from the field of chiropractics or physiotherapy. It is thought that the proper stabilization of this region of the body is crucial for coping with pain.

Therefore, the aim of the study was to assess the effectiveness of stabilizing training of deep core muscles in the lumbar spine in subjects in the age of 20-35 years, considering the progression level of degenerative disc disease: protrusion or extrusion, on the basis of the clinical condition.

ELIGIBILITY:
All the subjects undergo imaging examination in the form of MRI, whose results will be interpreted by a radiologist. Each person will be classified according to the current damage to the intervertebral disc as recommended by the American Society of Neuroradiology: protrusion or extrusion of the intervertebral disc.

Inclusion Criteria:

* disc disease located in the lumbar region of the spine confirmed by the MRI
* subacute stage of the disease
* age 20-35 years

Exclusion Criteria:

* advanced degenerative-deformatory changes of the spine
* previous fracture of the spine
* neurologic deficits in lower limbs or pelvis
* spondylolisthesis
* transitional vertebra
* rheumatic diseases

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
The Oswestry Disability Index | 15 minutes
  The Oswestry Disability Index (ODI) is a valid and reliable assessment tool used by clinicians and researchers to quantify disability for low back pain. The self-completed questionnaire contains ten sections concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. After completing, the score is calculated by by summing scores from all sections (total maximum points=50). Total results are calculated as a percentage. The higher the score, the subject's condition is worse.
  The results are interpreted as follows:
  0% to 20%: minimal disability 21%-40%: moderate disability 41%-60%: severe disability 61%-80%: crippled 81%-100%:These patients are either bed-bound or exaggerating their symptoms.
Range of motion evaluation | 15 minutes
  Range of motion will be evaluated SpinalMouse®. It is a non-invasive device used for assessing spinal mobility, whose reliability has been confirmed by studies. The measurement records the flexion and extension range of motion, and the test measure the total mobility from maximal flexion to maximal extension. Three measurements will be taken, and for statistical purposes their mean value will be calculated.

SECONDARY OUTCOMES:
The passive lumbar extension test | 10 minutes
  The passive lumbar extension test (PLE) is a tool for assessing the instability in the lumbar section of the spine. It is is the most suitable test for detecting lumbar instability, thanks to its excellent diagnostic accuracy, and good reliability
Straight leg raise test | 10 minutes
  Straight leg raise (SLR) test is considered by researchers to be sensitive and specific in diagnosing damage to the peripheral nervous system. The subject's lower limb with the knee extended was passively raised until potential symptoms were triggered, although not more than 60° of flexion in the hip joint, which, according to Kapandji, causes the maximum stretching of nerve structures.

CONTACTS AND LOCATIONS:
Overall Officials: Błażej Cieślik, PhD., Principal Investigator — University School of Physical Education, Wroclaw, Poland; Tomasz Kuligowski, PhD., Principal Investigator — University School of Physical Education, Wroclaw, Poland
Locations (1):
- theMedicine, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altinkaya N, Cekinmez M. Lumbar multifidus muscle changes in unilateral lumbar disc herniation using magnetic resonance imaging. Skeletal Radiol. 2016 Jan;45(1):73-7. doi: 10.1007/s00256-015-2252-z. Epub 2015 Sep 16. PMID 26377578
- [Background] Aluko A, DeSouza L, Peacock J. The effect of core stability exercises on variations in acceleration of trunk movement, pain, and disability during an episode of acute nonspecific low back pain: a pilot clinical trial. J Manipulative Physiol Ther. 2013 Oct;36(8):497-504.e1-3. doi: 10.1016/j.jmpt.2012.12.012. Epub 2013 Aug 12. PMID 23948426
- [Background] Leone A, Guglielmi G, Cassar-Pullicino VN, Bonomo L. Lumbar intervertebral instability: a review. Radiology. 2007 Oct;245(1):62-77. doi: 10.1148/radiol.2451051359. PMID 17885181
- [Background] Baek SO, Cho HK, Jung GS, Son SM, Cho YW, Ahn SH. Verification of an optimized stimulation point on the abdominal wall for transcutaneous neuromuscular electrical stimulation for activation of deep lumbar stabilizing muscles. Spine J. 2014 Sep 1;14(9):2178-83. doi: 10.1016/j.spinee.2014.02.016. Epub 2014 Feb 14. PMID 24534392
- [Background] Capra F, Vanti C, Donati R, Tombetti S, O'Reilly C, Pillastrini P. Validity of the straight-leg raise test for patients with sciatic pain with or without lumbar pain using magnetic resonance imaging results as a reference standard. J Manipulative Physiol Ther. 2011 May;34(4):231-8. doi: 10.1016/j.jmpt.2011.04.010. Epub 2011 May 5. PMID 21621724
- [Background] Dagenais S, Mayer J, Haldeman S, Borg-Stein J. Evidence-informed management of chronic low back pain with prolotherapy. Spine J. 2008 Jan-Feb;8(1):203-12. doi: 10.1016/j.spinee.2007.10.021. PMID 18164468
- [Background] Daghighi MH, Pouriesa M, Maleki M, Fouladi DF, Pezeshki MZ, Mazaheri Khameneh R, Bazzazi AM. Migration patterns of herniated disc fragments: a study on 1,020 patients with extruded lumbar disc herniation. Spine J. 2014 Sep 1;14(9):1970-7. doi: 10.1016/j.spinee.2013.11.056. Epub 2013 Dec 18. PMID 24361346